CLINICAL TRIAL: NCT00245024
Title: Phase IB Sulindac Study for Women at High Risk for Breast Cancer
Brief Title: Sulindac in Preventing Breast Cancer in Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: University of Arizona (Other)
Responsible Party: H. H. Sherry Chow, Arizona Cancer Center at University of Arizona Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000447144; P30CA023074 (NIH); UARIZ-UAZ04-2-02; UARIZ-HSC-0553
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ; lobular breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Sulindac

INTERVENTIONS:
Drug: sulindac
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of sulindac may prevent breast cancer.

PURPOSE: This randomized phase I trial is studying the effects of sulindac, to prevent breast cancer, in women at high risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the partitioning of sulindac and its metabolites in women at high risk for breast cancer by measuring drug and metabolite levels in nipple aspirate fluid (NAF) after 6 weeks of therapy.

Secondary

* Determine prostaglandin levels in the NAF of patients treated with this drug.
* Determine if NAG-1 levels are induced in the NAF of patients treated with this drug.
* Determine if C-reactive protein levels are reduced in the NAF of patients treated with this drug.
* Determine if NAG-1 levels and/or karyometric features in ductal epithelial cells are modulated in patients treated with this drug.

OUTLINE: This is a randomized, open-label study.

Patients undergo nipple aspirate fluid (NAF) collection. Patients are then randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sulindac once daily.
* Arm II: Patients receive oral sulindac twice daily. In both arms, treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. All patients then undergo a second NAF collection.

After completion of study treatment, patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 30 patients (15 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Gail assessment score > 1.7% risk for 5 years
  * History of lobular carcinoma in situ (pathology report required)
  * History of ductal carcinoma in situ (DCIS) (pathology report required)
  * History of breast cancer in ≥ 1 first-degree relative or history of BRCA1 or BRCA2 positivity not treated with oophorectomy or mastectomy (test report required)
  * History of breast cancer in ≥ 2 second-degree relatives
  * Any family history of breast cancer diagnosed prior to age 50
  * Personal history of breast cancer (invasive or DCIS) with 1 breast intact
* Nipple aspirate fluid production ≥ 5 microliters
* Negative mammogram for breast cancer within the past 10 months

  * Any suspicious breast masses must be examined by a clinical professional
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Pre- or postmenopausal

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No history of bleeding or clotting disorder

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.0 times upper limit of normal
* No indication of abnormal liver function

Renal

* Creatinine normal

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* No frequent, chronic, or moderate/severe gastric complaint
* No upper gastrointestinal problems (e.g., symptoms of heartburn, dyspepsia, or abdominal pain) requiring prescription or nonprescription medical remedies more than once per week (on average)
* No history of peptic ulcer or occult or gross intestinal bleeding

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction (e.g., urticaria, asthma, rhinitis) or gastric intolerance attributed to compounds of similar chemical or biological composition to sulindac
* No history of allergy attributed to lidocaine, EMLA® cream, or xylocaine
* No concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No more than 2-3 servings of alcohol per week during study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 6 months since prior chemotherapy for breast cancer (invasive or DCIS)

Endocrine therapy

* More than 6 months since prior hormonal therapy for breast cancer (invasive or DCIS)
* No concurrent hormone-suppressing agents (e.g., tamoxifen or anastrozole)
* No concurrent selective estrogen-receptor modulators
* No concurrent aromatase inhibitors

Radiotherapy

* More than 6 months since prior radiotherapy for breast cancer (invasive or DCIS)

Surgery

* See Disease Characteristics
* No prior breast duct-disrupting surgery (e.g., mastectomy) that would preclude ductoscopy

Other

* More than 3 months since prior warfarin or other systemic anticoagulant
* More than 4-6 weeks since prior nonsteroidal anti-inflammatory drugs
* No concurrent phenytoin or sulfonamides
* No concurrent warfarin or other systemic anticoagulant
* No other concurrent nonsteroidal anti-inflammatory drugs (including low-dose aspirin)
* No concurrent large doses of supplements, vitamins (> regular daily multivitamin) and/or herbal medicines (e.g., echinacea, ginkgo biloba, Hypericum perforatum [St. John's wort], or herbal tea)
* No other concurrent investigational agents

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Sulindac and sulindac metabolite levels in nipple aspirate fluid (NAF) after 6 weeks of treatment

SECONDARY OUTCOMES:
Prostaglandin (PGE2) levels in NAF before and after 6 weeks of treatment
NAG-1 induction and C-reactive protein (CRP) reduction before and after 6 weeks of treatment
Magnitude of change and dose response of PGE2, NAG-1, and CRP in NAF before and after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Thompson, PhD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Thompson PA, Huang C, Yang J, Wertheim BC, Roe D, Zhang X, Ding J, Chalasani P, Preece C, Martinez J, Chow HS, Stopeck AT. Sulindac, a Nonselective NSAID, Reduces Breast Density in Postmenopausal Women with Breast Cancer Treated with Aromatase Inhibitors. Clin Cancer Res. 2021 Oct 15;27(20):5660-5668. doi: 10.1158/1078-0432.CCR-21-0732. Epub 2021 Jun 10. PMID 34112707